CLINICAL TRIAL: NCT01814553
Title: A Phase IIIb, Non-randomized, Open-label, Two-cohort Study in Patients With EGFR Mutations-positive Advanced Adenocarcinoma of the Lung, Assessing the Utility of the Afatinib Diarrhea Assessment and Management Guidelines (ADAM)
Brief Title: ADAM-Afatinib Diarrhea Assessment and Management
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1200.167
Record Dates: First submitted 2013-03-04; First posted 2013-03-20 (Estimated); Results first posted 2016-10-31 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-09

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; Loperamide

ARMS (2):
- Afatinib 40 mg + Loperamide (Cohort 1) (Experimental): afatinib starting 40 mg daily; Cohort 1 will receive loperamide at first sign of diarrhea; Cohort 2 will receive loperamide starting C1D1.
  Interventions: Drug: afatinib; Drug: loperamide
- Afatinib 40 mg + loperamide prophylactic (Cohort 2) (Experimental): afatinib starting 40 mg daily; Cohort 1 will receive loperamide at first sign of diarrhea; Cohort 2 will receive loperamide starting C1D1.
  Interventions: Drug: afatinib; Drug: loperamide

INTERVENTIONS:
Drug: afatinib — Daily treatment starting 40 mg per day
Drug: loperamide — Follow cohort assignment and diarrhea management guidelines

SUMMARY:
This is a non-randomized, open label, two-cohort, multi-institutional study to evaluate the use of diarrheal management tools intended to facilitate timely intervention and treatment modifications due to afatinib treatment-related diarrhea in patients with EGFR mutations-positive adenocarcinoma of the lung. Patients in Cohort 1 will follow diarrhea management. Patients in Cohort 2 will receive prophylactic loperamide starting the fist day of afatinib treatment.

ELIGIBILITY:
Inclusion criteria:

1. Pathologically confirmed diagnosis of Stage IIIB or Stage IV adenocarcinoma of the lung, with EGFR mutations-positive status, who are not eligible to receive surgery or chemoradiotherapy. Patients with mixed histology are eligible if adenocarcinoma is the predominant histology, and is a suitable candidate for EGFR-TKI monotherapy, in the opinion of the investigator.
2. Patients must have Epidermal Growth Factor Receptor (EGFR) mutation-positive status according to the institutional standard of care.
3. Patient received no more than one (1) prior chemotherapy for locally advanced or metastatic adenocarcinoma of the lung.
4. Male or female patients Age 18 years and older.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
6. Adequate organ function, defined as all of the following:

   * Left Ventricular Ejection Fraction (LVEF) of above 50% or within institution normal values
   * Absolute neutrophil count (ANC) above 1500 / mm3.
   * Platelet count above 75,000 / mm3.
   * Estimated creatinine clearance more than 45ml / min.
   * Total Bilirubin less than 1.5 times upper limit of (institutional/central) normal
   * Aspartate amino transferase (AST) or alanine amino transferase (ALT) less than three times the upper limit of (institutional/central) normal (ULN) (if related to liver metastases less than five times ULN).
7. Recovered from any previous therapy related toxicity to Grade 0 or 1 at study entry
8. Able and willing to follow diarrhea management guidelines provided under this study and to complete Diarrhea Management Worksheet as instructed.

Exclusion criteria:

1. Chemotherapy, biological therapy or investigational agents within four weeks prior to the start of study treatment.
2. Prior treatment with EGFR directed small molecules or antibodies.
3. Hormonal treatment within 2 weeks prior to start of study treatment (continued use of anti-androgens and/or gonadorelin analogues for treatment of prostate cancer permitted).
4. Major surgery within 4 weeks before starting study treatment or scheduled for surgery during the projected course of the study.
5. Known hypersensitivity to afatinib or the excipients of any of the trial drugs.
6. History or presence of clinically relevant cardiovascular abnormalities.
7. Any history of or concomitant condition that, in the opinion of the Investigator, would compromise the patient¿s ability to comply with the study or interfere with the evaluation of the efficacy and safety of the test drug.
8. Previous or concomitant invasive malignancies at other sites.
9. Known pre-existing interstitial lung disease (ILD).
10. Any history or presence of poorly controlled gastrointestinal disorders that could affect the absorption of the study drug.

14. Active hepatitis B infection, active hepatitis C infection and/or known HIV carrier, who are determined by the investigator as not a suitable candidate to receive EGFR-TKI treatment.

15. Patients with meningeal carcinomatosis. 16. Patients with brain or subdural metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (12):
- United States (12):
  - 1200.167.01009 Boehringer Ingelheim Investigational Site, Santa Rosa, California
  - 1200.167.01020 Boehringer Ingelheim Investigational Site, Orlando, Florida
  - 1200.167.01018 Boehringer Ingelheim Investigational Site, Port Saint Lucie, Florida
  - 1200.167.01012 Boehringer Ingelheim Investigational Site, St. Petersburg, Florida
  - 1200.167.01007 Boehringer Ingelheim Investigational Site, Skokie, Illinois
  - 1200.167.01008 Boehringer Ingelheim Investigational Site, Skokie, Illinois
  - 1200.167.01001 Boehringer Ingelheim Investigational Site, Morristown, New Jersey
  - 1200.167.01014 Boehringer Ingelheim Investigational Site, Corvallis, Oregon
  - 1200.167.01002 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 1200.167.01006 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 1200.167.01005 Boehringer Ingelheim Investigational Site, Nashville, Tennessee
  - 1200.167.01003 Boehringer Ingelheim Investigational Site, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: PD: Progressive Disease (PD)
Groups:
- Afatinib 40 mg + Loperamide (Cohort 1): Subjects were orally administered with the starting dose of Afatinib Film-coated tablets 40 mg once daily - with possible dose reductions to 30 mg and 20 mg and if any diarrhea was experienced Common Terminology Criteria for Adverse Events (CTCAE Grade 1), 2 tablets of loperamide 2 mg were to be taken immediately, followed by 1 tablet of loperamide 2 mg with every subsequent loose bowel movement until bowel movements ceased for 12 hours.
- Afatinib 40 mg + Loperamide Prophylactic (Cohort 2): Subjects were orally administered with the starting dose of Afatinib Film-coated tablets 40 mg once daily - with possible dose reductions to 30 mg and 20 mg and 2 tablets of loperamide 2 mg daily (i.e., 4 mg daily) starting on Course 1 Day 1. If any diarrhea was experienced (CTCAE Grade 1) by subjects, 2 tablets of loperamide 2 mg were to be taken immediately, followed by 1 tablet of loperamide 2mg with every subsequent loose bowel movement until bowel movements ceased for 12 hours. Subjects who experienced no diarrhea during Course 1 were allowed to reduce the loperamide dose to 2 mg daily and subjects who experienced no diarrhea during the first two courses discontinued daily prophylactic loperamide at the end of Course 2.
Period: Overall Study
Arm/Group | Afatinib 40 mg + Loperamide (Cohort 1) | Afatinib 40 mg + Loperamide Prophylactic (Cohort 2)
Started | 18 | 22
Completed | 0 | 0
Not Completed | 18 | 22
Not completed — PD per clinical progression | 6 | 8
Not completed — Other Adverse Event | 4 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Other than stated | 7 | 8

BASELINE CHARACTERISTICS:
Population: Treated Set : This analysis set includes all entered patients who received at least one dose of investigational treatment (afatinib) and for whom there was documentation that they took at least 1 dose.
Groups:
- Total: Total of all reporting groups
Arm/Group | Afatinib 40 mg + Loperamide (Cohort 1) | Afatinib 40 mg + Loperamide Prophylactic (Cohort 2) | Total
Number analyzed (Participants) | 18 | 22 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.70 (10.80) | 68.00 (6.50) | 68.80 (8.62)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 6 | 10 | 16

OUTCOME MEASURES:

1. Primary Outcome: Occurence of CTCAE Grade >= 2 Diarrhea
Description: Overall incidence of patients who experienced diarrhea during the first three courses of afatinib treatment.
Time Frame: From first drug administration until 28 days after the end of third treatment course, up to 84 days.
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib 40 mg + Loperamide (Cohort 1) | Afatinib 40 mg + Loperamide Prophylactic (Cohort 2)
Number analyzed (Participants) | 18 | 22
Percentage of participants | 72.20 | 31.80

2. Secondary Outcome: Time to Initial Onset of Diarrhea Grade 2 or Higher
Description: Time to initial onset of diarrhea grade 2 or higher
Time Frame: From first drug administration until end of third treatment course, up to 84 days.
Population: Treated set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Afatinib 40 mg + Loperamide (Cohort 1) | Afatinib 40 mg + Loperamide Prophylactic (Cohort 2)
Number analyzed (Participants) | 13 | 7
days | 23.50 (22.64) | 15.40 (14.97)

3. Secondary Outcome: Duration of First Episode of Diarrhea Grade 2 or Higher
Description: Duration of first episode of diarrhea grade 2 or higher.
  Please note that the nine patients experienced diarrhea episodes that were not managed according to the protocol specified afatinib treatment interruptions and dose reductions. No patients were excluded from the primary analysis.
Time Frame: From first drug administration until end of third treatment course, up to 84 days.
Population: Treated set
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Afatinib 40 mg + Loperamide (Cohort 1) | Afatinib 40 mg + Loperamide Prophylactic (Cohort 2)
Number analyzed (Participants) | 13 | 7
days | 3.10 (4.09) | 7.60 (5.19)

4. Secondary Outcome: Changes in Intensity of Diarrhea Over Time
Description: Percentage of participants with grade 2 or higher diarrhea each week for the first 3 cycles of afatinib treatment
Time Frame: Up to 12 weeks (equivalent to 3 courses)
Population: Treated set
Measure: Number; unit: Percentage of participants
Arm/Group | Afatinib 40 mg + Loperamide (Cohort 1) | Afatinib 40 mg + Loperamide Prophylactic (Cohort 2)
Number analyzed (Participants) | 18 | 22
Percentage of participants
  Grade 2: Week 1 (N=2, 1) | 11.10 | 4.50
  Grade 2: Week 2 (N=4, 3) | 22.20 | 13.60
  Grade 2: Week 3 (N=3, 3) | 16.70 | 13.60
  Grade 2: Week 4 (N=6, 2) | 33.30 | 9.10
  Grade 2: Week 5 (N=2, 0) | 11.10 | 0.00
  Grade 2: Week 6 (N=0, 1) | 0.00 | 4.80
  Grade 2: Week 7 (N=2, 1) | 11.80 | 5.00
  Grade 2: Week 8 (N=3, 0) | 17.60 | 0.00
  Grade 2: Week 9 (N=2, 0) | 11.80 | 0.00
  Grade 2: Week 10 (N=0, 0) | 0.00 | 0.00
  Grade 2: Week 11 (N=2, 0) | 11.80 | 0.00
  Grade 2: Week 12 (N=1, 1) | 5.90 | 6.30
  Grade >=3: Week 1 (N=1, 1) | 5.60 | 4.50
  Grade >=3: Week 2 (N=2, 2) | 11.10 | 9.10
  Grade >=3: Week 3 (N=3, 1) | 16.70 | 4.50
  Grade >=3: Week 4 (N=0, 1) | 0.00 | 4.50
  Grade >=3: Week 5 (N=0, 0) | 0.00 | 0.00
  Grade >=3: Week 6 (N=0, 0) | 0.00 | 0.00
  Grade >=3: Week 7 (N=1, 0) | 5.90 | 0.00
  Grade >=3: Week 8 (N=0, 0) | 0.00 | 0.00
  Grade >=3: Week 9 (N=0, 0) | 0.00 | 0.00
  Grade >=3: Week 10 (N=1, 0) | 5.90 | 0.00
  Grade >=3: Week 11 (N=0, 0) | 0.00 | 0.00
  Grade >=3: Week 12 (N=0, 0) | 0.00 | 0.00

5. Secondary Outcome: PFS
Description: Progression-free survival (PFS). PFS was defined as the time from the start of treatment to an event occurred. In the analyses for the PFS endpoint, an event was defined as disease progression or death, whichever occurred earlier. Data for patients who did not die or progress during the trial were censored at the time of afatinib discontinuation or transition to commercially available afatinib. Median PFS is estimated using Kaplan-Meier method.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1).
Time Frame: Every 08 weeks during the first 6 months of treatment, and every 12 weeks thereafter until the end of treatment.
Population: Treated Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Afatinib 40 mg + Loperamide (Cohort 1) | Afatinib 40 mg + Loperamide Prophylactic (Cohort 2)
Number analyzed (Participants) | 18 | 22
Months | 15.40 [5.50 to NA] — The upper limit was not evaluable due to insufficient patients. | 9.90 [5.50 to NA] — The upper limit was not evaluable due to insufficient patients.

ADVERSE EVENTS:
Time Frame: From first drug administration until 28 days after the end of third treatment course, up to 112 days.
Arm/Group | Afatinib 40 mg + Loperamide (Cohort 1) | Afatinib 40 mg + Loperamide Prophylactic (Cohort 2)
Serious Adverse Events (participants affected / at risk) | 10/18 | 5/22
Other Adverse Events (participants affected / at risk) | 18/18 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg + Loperamide (Cohort 1) (N=18) | Afatinib 40 mg + Loperamide Prophylactic (Cohort 2) (N=22)
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Abscess limb (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 40 mg + Loperamide (Cohort 1) (N=18) | Afatinib 40 mg + Loperamide Prophylactic (Cohort 2) (N=22)
Anaemia (Blood and lymphatic system disorders) | 5 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Diplopia (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 2 | 0
Eyelash hyperpigmentation (Eye disorders) | 1 | 0
Eyelid irritation (Eye disorders) | 1 | 0
Eyelid rash (Eye disorders) | 1 | 0
Growth of eyelashes (Eye disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 2
Macular degeneration (Eye disorders) | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Chapped lips (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 11
Defaecation urgency (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 16 | 18
Dry mouth (Gastrointestinal disorders) | 0 | 3
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 2
Frequent bowel movements (Gastrointestinal disorders) | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Lip blister (Gastrointestinal disorders) | 1 | 0
Lip dry (Gastrointestinal disorders) | 2 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 12 | 8
Retching (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 7 | 6
Vomiting (Gastrointestinal disorders) | 3 | 3
Asthenia (General disorders) | 2 | 0
Chest pain (General disorders) | 1 | 0
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 8 | 5
Gait disturbance (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 8 | 3
Non-cardiac chest pain (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 4 | 1
Pyrexia (General disorders) | 2 | 0
Xerosis (General disorders) | 1 | 2
Candida infection (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 1 | 0
Nail infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 1 | 0
Rash pustular (Infections and infestations) | 0 | 2
Rhinitis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 4 | 2
Wound infection (Infections and infestations) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 1
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Blood magnesium decreased (Investigations) | 2 | 0
Blood phosphorus decreased (Investigations) | 2 | 0
Weight decreased (Investigations) | 5 | 2
Decreased appetite (Metabolism and nutrition disorders) | 7 | 4
Dehydration (Metabolism and nutrition disorders) | 7 | 5
Gout (Metabolism and nutrition disorders) | 0 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 2
Dysgeusia (Nervous system disorders) | 4 | 4
Headache (Nervous system disorders) | 3 | 1
Lethargy (Nervous system disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 2 | 0
Neuropathy peripheral (Nervous system disorders) | 2 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 3
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Nasal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal ulcer (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 7 | 8
Dry skin (Skin and subcutaneous tissue disorders) | 8 | 4
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hair growth abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 1
Nail toxicity (Skin and subcutaneous tissue disorders) | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 3 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 2 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3
Rash (Skin and subcutaneous tissue disorders) | 7 | 4
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 1 | 3
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flush (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
In this study, Nine patients experienced diarrhea episodes that were not managed according to the protocol specified afatinib treatment interruptions and dose reductions. No patients were excluded from the primary analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.